CLINICAL TRIAL: NCT04113148
Title: Optical Pressure Ulcer Study: Tissue Vascular Optics and Impedance Measurements for the Detection of Early Tissue Damage and Pressure Ulceration
Brief Title: Tissue Vascular Optics and Impedance Measurements for the Detection of Early Tissue Damage and Pressure Ulceration
Acronym: OPUS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: FO18022; 8779 (Other: The Newcastle upon Tyne Hospitals NHS FT)
Record Dates: First submitted 2019-07-04; First posted 2019-10-02 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-10

CONDITIONS: Pressure Ulcer
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Healthy volunteer: Physiological measurements from heel over 60 minute period
  Interventions: Other: Physiological measurements from heel
- At risk of Pressure Ulcer: Physiological measurements from heel over 60 minute period
  Interventions: Other: Physiological measurements from heel
- Confirmed Catefory I Pressure Ulcer: Physiological measurements from heel over 60 minute period
  Interventions: Other: Physiological measurements from heel
- Suspected Deep Tissue Injury: Physiological measurements from heel over 60 minute period
  Interventions: Other: Physiological measurements from heel

INTERVENTIONS:
Other: Physiological measurements from heel — Measurements of blood flow, tissue oxygen saturation, temperature, pressure

SUMMARY:
Pressure ulcers are common, distressing and expensive. Currently scoring systems and checks by nursing staff are carried out to assess a patient's risk of developing a pressure ulcer.

The investigators would like to see whether non-invasive measurements can be taken from patients to predict who might be at risk of pressure ulcers to allow us to intervene and reduce the risk of it happening.

DETAILED DESCRIPTION:
Pressure ulcers are common, distressing and expensive. Currently scoring systems and checks by nursing staff are carried out to assess a patient's risk of developing a pressure ulcer.

The aim is to investigate whether non-invasive physiological measurements can be taken from patients to predict who might be at risk of pressure ulcers to allow us to intervene and reduce the risk.

ELIGIBILITY:
Inclusion Criteria:

HEALTHY VOLUNTEERS:

* Able to give consent
* Male or female
* Over the age of 18 years
* No known peripheral vascular disease
* No known tissue damage
* Able to read and understand basic English language

PATIENTS:

* Able to give consent
* Male or female
* Over the age of 18 years
* Either at risk (Braden scale <17) or confirmed Category 1 or 2 PU or confirmed DTI
* Well enough to attend lab without any attachments (IV fluids, IV medications, oxygen)
* Able to transfer to bed with assistance of one
* Able to read and understand basic English Language

Exclusion Criteria:

HEALTHY VOLUNTEERS:

* Presence of tissue damage or ulceration in the foot
* Known peripheral vascular disease
* Known hypersensitivity to fixation tape
* Presence of a pacemaker
* Participants unable to or refusing to give informed consent

PATIENTS:

* Known hypersensitivity to fixation tape
* Participants unable to or refusing to give informed consent
* Unable to transfer to bed with assistance of one.
* Requiring more than routine observations and requiring attachments (IV fluids, IV medications, oxygen)
* Presence of a pacemaker

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: From in patient population
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-11 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Laser Doppler Flowmetry | 20 minutes
  Laser light to assess perfusion of heel
Spectrometry | 20 minutes
  Light spectrometry to assess tissue oxygen saturation of the heel
Impedance | 5 minutes
  Measurement of oedema of the heel
Temperature | 5 minutes
  Thermal image of heel to assess skin temperature

SECONDARY OUTCOMES:
Co-morbidities | 5 minutes
  The presence of peripheral arterial disease, ischaemic heart disease, diabetes and previous pressure ulcers

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Stansby, MBBS, Principal Investigator — Newcastle upon Tyne NHS Hospitals Foundation Trust/Newcastle University
Locations (1):
- Vascular Dept, Newcastle, Tyne and Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Data is anonymised